CLINICAL TRIAL: NCT04662619
Title: A Proof-of-Concept, Randomized, Double-Blind, Placebo-Controlled, Two-Arm, Parallel-Group, Nutritional Intervention Study to Examine the Clinical and Immunological Effects of a Probiotic Food Supplement Containing B. Infantis (EVC001) in Healthy Breastfed Infants at Risk of Developing Atopic Dermatitis
Brief Title: A Study of a Probiotic Food Supplement Containing B. Infantis (EVC001) in Healthy Breastfed Infants at Risk of Developing Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Collaborators: Infinant Health, Inc. (formerly known as Evolve BioSystems, Inc.) (Unknown)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CCSNUT002443; CCSNUT002443 (Other: Johnson & Johnson Consumer Inc.)
Record Dates: First submitted 2020-11-26; First posted 2020-12-10 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B. infantis (Experimental): A once-daily feeding of activated B. infantis EVC001 (8.0 *10^9 colony forming units [CFU]) will be provided to infants for 12 weeks.
  Interventions: Other: B. infantis
- Placebo (Placebo Comparator): A once-daily oral feeding of lactose placebo will be provided to infants for 12 weeks.
  Interventions: Other: Lactose Placebo

INTERVENTIONS:
Other: B. infantis — Bifidobacterium longum subspecies infantis strain EVC001, designated a "Foods for Special Dietary Use" (FSDU), will be provided to infants once daily for 12 weeks.
  Other Names: Evivo
  Arms: B. infantis
Other: Lactose Placebo — Powdered infant formula grade lactose will be provided to infants once daily for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of B. infantis (EVC001) versus placebo supplementation, in healthy breastfed infants at risk of developing atopic dermatitis (AD), on cumulative incidence of physician-diagnosed AD during the first year of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infant
* Has at least one first degree relative (that is biological parent or full sibling) with a history of atopic disease (that is mother-reported, physician-diagnosed Atopic Dermatitis (AD), allergic rhinitis, or asthma)
* Breastfeeding established (as determined by the principal Investigator [PI] or designee) at the time of study enrollment (Day 0), with maternal intent to maintain exclusive breastfeeding for greater than or equal to (>=)12 weeks
* Will participate in the study under supervision of his/her biological mother ("Caregiver") who is: a) At least 18 years old b) The legal guardian of the infant c) Intending to cohabitate with the infant for the duration of the study d) Willing to follow all Caregiver responsibilities e) Fluent in Finnish, Swedish, or English
* The PI considers the Caregiver likely to adequately comply with the study protocol requirements based on demonstrated compliance with antenatal appointments and agreement to complete the intuitive, interactive, electronic diary (eDiary) utilizing personal smart device (example, tablet, cell phone)

Exclusion Criteria:

* Preterm delivery (< 36 weeks [252 days] gestational age)
* Admission to the neonatal unit for issues other than establishment of normal feeding
* Evidence of a baseline illness/condition (example abnormal birth weight) or significant risk of developing an illness/condition (based on review of maternal/pregnancy information) that would, in the opinion of the Principal Investigator (PI) or designee, introduce a significant safety concern if the infant were enrolled in the study or otherwise preclude study participation
* Significant birth defect/complication that would, in the opinion of the PI or designee, create a safety concern or otherwise confound the study (example, abdominal wall defects, congenital heart disease)
* Severe widespread skin condition (example collodion)
* Has consumed greater than (>)100 milliliter (mL) of formula per day within the 48 hours prior to enrollment (Day 0)
* Twin or multiple births
* Atopic dermatitis (AD) diagnosed at Day 0
* Has a history of confirmed coronavirus disease 2019 (COVID-19) within 30 days prior to any on-site visit
* Within 14 days prior to Visit 1, has been in close contact (exposure within 6 feet for a cumulative time of 15 minutes or more over a 24-hour period) with anyone who has a confirmed case of COVID-19
* Is under a COVID-19 isolation/quarantine order
* Has had self-reported (for Caregiver) or parent-reported (for infant) symptoms of COVID-19 within 14 days prior to the screening visit, such as unexplained cough, shortness of breath/difficulty breathing, fatigue, body aches (headaches, muscle pain, stomachaches), conjunctivitis, loss of smell, loss of taste, poor appetite, nausea, vomiting, diarrhea, palpitations, or chest pain/tightness

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 273 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Atopic Dermatitis (AD) through Week 52 | Up to Week 52
  Percentage of participants with atopic dermatitis (AD) through Week 52 will be reported. AD will be diagnosed if three of the following four criteria are met: 1) pruritus, 2) typical morphology and distribution (facial and extensor involvement), 3) chronic or chronically relapsing dermatitis, 4) personal or family history of atopic disease.

SECONDARY OUTCOMES:
Percentage of Infants with Adverse Events Through Weeks 12, 52 and 104 | Up to Weeks 12, 52 and 104
  The percentage of infants with AEs, serious adverse events (SAEs), AEs leading to discontinuation, and AEs related to the gastrointestinal system will be determined at Weeks 12, 52 and 104.
Percentage of Participants with Atopic Dermatitis (AD) Through Weeks 24 and 104 | Up to Weeks 24 and 104
  Percentage of participants with AD through Week 24 and 104 will be reported. AD will be diagnosed if three of the following four criteria are met: 1) pruritus, 2) typical morphology and distribution (facial and extensor involvement), 3) chronic or chronically relapsing dermatitis, 4) personal or family history of atopic disease.
Time to Onset of AD Through Weeks 52 and 104 | Up to Weeks 52 and 104
  Time to onset of AD through Weeks 52 and 104 will be reported.
Percentage of Infants with B. infantis Gut Colonization at Week 12 | Week 12
  Percentage of infants with B. infantis gut colonization at Week 12 will be reported.
Percentage of Participants with at least Mild Atopic Dermatitis (AD) Severity Based on the Eczema Area and Severity Index (EASI) Score at Weeks 12, 52, and 104 | At Weeks 12, 52, and 104
  Percentage of participants with at least mild Atopic Dermatitis (AD) severity based on the EASI score at Weeks 12, 52, and 104 will be reported. Physician rates severity of four parameters: erythema, infiltration, excoriation and lichenification on a scale of 0 (none) to 3 (severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Physician determines how much area is affected on a scale of 0 (none) to 6 (90 to 100%). A body region score is determined by multiplying the sum of the severity scores by the affected area score by a constant corresponding to the relative body surface area for that body region (20%, 30%, 20%, and 30%, respectively). The 4 body region scores are summed to yield the EASI score which ranges from 0 to 72, with a higher score indicating more severe AD. The AD onset in the study's population can be diagnosed throughout the study at either scheduled or unscheduled visits starting as early as 1 month of age.
Time to Onset of at least Mild Atopic Dermatitis (AD) Severity Based on the Eczema Area and Severity Index (EASI) Score | At the time of AD onset (up to Week 104)
  Time to onset of at least mild Atopic Dermatitis (AD) severity based on the EASI score up to Week 104 will be reported. Physician rates severity of four parameters: erythema, infiltration, excoriation and lichenification on a scale of 0 (none) to 3 (severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Physician determines how much area is affected on a scale of 0 (none) to 6 (90 to 100%). A body region score is determined by multiplying the sum of the severity scores by the affected area score by a constant corresponding to the relative body surface area for that body region (20%, 30%, 20%, and 30%, respectively). The 4 body region scores are summed to yield the EASI score which ranges from 0 to 72, with a higher score indicating more severe AD. The AD onset in the study's population can be diagnosed throughout the study at either scheduled or unscheduled visits starting as early as 1 month of age.
Percentage of Participants with at least Mild AD Severity Based on the Patient-Oriented Eczema Measure (POEM) Score at Weeks 12, 52, and 104 | At Weeks 12, 52, and 104
  The POEM is a simple, valid, easily interpreted, and reproducible tool for assessing AD and monitoring aspects of the disease that are important to participants with AD. Study Personnel will interview Caregivers at time of AD diagnosis and (only for participants with AD) at Weeks 12, 52, and 104 to rate seven symptoms (itchy skin, sleep disturbance, bleeding skin, skin weeping/oozing, skin flaking, skin cracking, skin dryness/roughness) using a 5-point scale of frequency of occurrence during the previous week (no days, 1-2 days, 3-4 days, 5-6 days, every day). The total score is the sum of the 7 items which is ranged from 0 to 28; a high score is indicative of more severe AD. The AD onset in the study's population can be diagnosed throughout the study at either scheduled or unscheduled visits starting as early as 1 month of age.
Time to Onset of at least Mild AD Severity Based on the Patient-Oriented Eczema Measure (POEM) Score | At the time of AD onset (up to Week 104)
  The POEM is a simple, valid, easily interpreted, and reproducible tool for assessing AD and monitoring aspects of the disease that are important to participants with AD. Study Personnel will interview Caregivers at time of AD diagnosis and (only for participants with AD) at Weeks 12, 52, and 104 to rate seven symptoms (itchy skin, sleep disturbance, bleeding skin, skin weeping/oozing, skin flaking, skin cracking, skin dryness/roughness) using a 5-point scale of frequency of occurrence during the previous week (no days, 1-2 days, 3-4 days, 5-6 days, every day). The total score is the sum of the 7 items which is ranged from 0 to 28; a high score is indicative of more severe AD. The AD onset in the study's population can be diagnosed throughout the study at either scheduled or unscheduled visits starting as early as 1 month of age.

CONTACTS AND LOCATIONS:
Overall Officials: Samuli Rautava, M.D., Ph.D., Principal Investigator — Helsinki University Central Hospital
Locations (1):
- HUS Children and Adolescents, Clinical Trial Unit, Park Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrahamsson TR, Jakobsson HE, Andersson AF, Bjorksten B, Engstrand L, Jenmalm MC. Low diversity of the gut microbiota in infants with atopic eczema. J Allergy Clin Immunol. 2012 Feb;129(2):434-40, 440.e1-2. doi: 10.1016/j.jaci.2011.10.025. Epub 2011 Dec 6. PMID 22153774
- [Background] Abrahamsson TR, Jakobsson T, Bottcher MF, Fredrikson M, Jenmalm MC, Bjorksten B, Oldaeus G. Probiotics in prevention of IgE-associated eczema: a double-blind, randomized, placebo-controlled trial. J Allergy Clin Immunol. 2007 May;119(5):1174-80. doi: 10.1016/j.jaci.2007.01.007. Epub 2007 Mar 8. PMID 17349686
- [Background] Allen KJ, Remington BC, Baumert JL, Crevel RW, Houben GF, Brooke-Taylor S, Kruizinga AG, Taylor SL. Allergen reference doses for precautionary labeling (VITAL 2.0): clinical implications. J Allergy Clin Immunol. 2014 Jan;133(1):156-64. doi: 10.1016/j.jaci.2013.06.042. Epub 2013 Aug 26. PMID 23987796
- [Background] Belkaid Y, Harrison OJ. Homeostatic Immunity and the Microbiota. Immunity. 2017 Apr 18;46(4):562-576. doi: 10.1016/j.immuni.2017.04.008. PMID 28423337
- [Background] Cabana MD, McKean M, Caughey AB, Fong L, Lynch S, Wong A, Leong R, Boushey HA, Hilton JF. Early Probiotic Supplementation for Eczema and Asthma Prevention: A Randomized Controlled Trial. Pediatrics. 2017 Sep;140(3):e20163000. doi: 10.1542/peds.2016-3000. Epub 2017 Aug 7. PMID 28784701
- [Background] Casaburi G, Duar RM, Vance DP, Mitchell R, Contreras L, Frese SA, Smilowitz JT, Underwood MA. Early-life gut microbiome modulation reduces the abundance of antibiotic-resistant bacteria. Antimicrob Resist Infect Control. 2019 Aug 14;8:131. doi: 10.1186/s13756-019-0583-6. eCollection 2019. PMID 31423298
- [Background] Charman CR, Venn AJ, Williams HC. The patient-oriented eczema measure: development and initial validation of a new tool for measuring atopic eczema severity from the patients' perspective. Arch Dermatol. 2004 Dec;140(12):1513-9. doi: 10.1001/archderm.140.12.1513. PMID 15611432
- [Background] Charman CR, Venn AJ, Ravenscroft JC, Williams HC. Translating Patient-Oriented Eczema Measure (POEM) scores into clinical practice by suggesting severity strata derived using anchor-based methods. Br J Dermatol. 2013 Dec;169(6):1326-32. doi: 10.1111/bjd.12590. PMID 24024631
- [Background] Chiu CY, Yang CH, Su KW, Tsai MH, Hua MC, Liao SL, Lai SH, Chen LC, Yeh KW, Huang JL. Early-onset eczema is associated with increased milk sensitization and risk of rhinitis and asthma in early childhood. J Microbiol Immunol Infect. 2020 Dec;53(6):1008-1013. doi: 10.1016/j.jmii.2019.04.007. Epub 2019 May 8. PMID 31129013
- [Background] Cuello-Garcia CA, Brozek JL, Fiocchi A, Pawankar R, Yepes-Nunez JJ, Terracciano L, Gandhi S, Agarwal A, Zhang Y, Schunemann HJ. Probiotics for the prevention of allergy: A systematic review and meta-analysis of randomized controlled trials. J Allergy Clin Immunol. 2015 Oct;136(4):952-61. doi: 10.1016/j.jaci.2015.04.031. Epub 2015 Jun 2. PMID 26044853
- [Background] Fiocchi A, Pawankar R, Cuello-Garcia C, Ahn K, Al-Hammadi S, Agarwal A, Beyer K, Burks W, Canonica GW, Ebisawa M, Gandhi S, Kamenwa R, Lee BW, Li H, Prescott S, Riva JJ, Rosenwasser L, Sampson H, Spigler M, Terracciano L, Vereda-Ortiz A, Waserman S, Yepes-Nunez JJ, Brozek JL, Schunemann HJ. World Allergy Organization-McMaster University Guidelines for Allergic Disease Prevention (GLAD-P): Probiotics. World Allergy Organ J. 2015 Jan 27;8(1):4. doi: 10.1186/s40413-015-0055-2. eCollection 2015. PMID 25628773
- [Background] Foolad N, Brezinski EA, Chase EP, Armstrong AW. Effect of nutrient supplementation on atopic dermatitis in children: a systematic review of probiotics, prebiotics, formula, and fatty acids. JAMA Dermatol. 2013 Mar;149(3):350-5. doi: 10.1001/jamadermatol.2013.1495. PMID 23682371
- [Background] Frese SA, Hutton AA, Contreras LN, Shaw CA, Palumbo MC, Casaburi G, Xu G, Davis JCC, Lebrilla CB, Henrick BM, Freeman SL, Barile D, German JB, Mills DA, Smilowitz JT, Underwood MA. Persistence of Supplemented Bifidobacterium longum subsp. infantis EVC001 in Breastfed Infants. mSphere. 2017 Dec 6;2(6):e00501-17. doi: 10.1128/mSphere.00501-17. eCollection 2017 Nov-Dec. PMID 29242832
- [Background] Ganemo A, Svensson A, Svedman C, Gronberg BM, Johansson AC, Wahlgren CF. Usefulness of Rajka & Langeland Eczema Severity Score in Clinical Practice. Acta Derm Venereol. 2016 May;96(4):521-4. doi: 10.2340/00015555-2302. PMID 26611655
- [Background] Gensollen T, Iyer SS, Kasper DL, Blumberg RS. How colonization by microbiota in early life shapes the immune system. Science. 2016 Apr 29;352(6285):539-44. doi: 10.1126/science.aad9378. PMID 27126036
- [Background] Hanifin JM, Thurston M, Omoto M, Cherill R, Tofte SJ, Graeber M. The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. EASI Evaluator Group. Exp Dermatol. 2001 Feb;10(1):11-8. doi: 10.1034/j.1600-0625.2001.100102.x. PMID 11168575
- [Background] Henrick BM, Hutton AA, Palumbo MC, Casaburi G, Mitchell RD, Underwood MA, Smilowitz JT, Frese SA. Elevated Fecal pH Indicates a Profound Change in the Breastfed Infant Gut Microbiome Due to Reduction of Bifidobacterium over the Past Century. mSphere. 2018 Mar 7;3(2):e00041-18. doi: 10.1128/mSphere.00041-18. eCollection 2018 Mar-Apr. PMID 29564397
- [Background] Henrick BM, Chew S, Casaburi G, Brown HK, Frese SA, Zhou Y, Underwood MA, Smilowitz JT. Colonization by B. infantis EVC001 modulates enteric inflammation in exclusively breastfed infants. Pediatr Res. 2019 Dec;86(6):749-757. doi: 10.1038/s41390-019-0533-2. Epub 2019 Aug 23. PMID 31443102
- [Background] Hooper LV, Littman DR, Macpherson AJ. Interactions between the microbiota and the immune system. Science. 2012 Jun 8;336(6086):1268-73. doi: 10.1126/science.1223490. Epub 2012 Jun 6. PMID 22674334
- [Background] Isolauri E, Arvola T, Sutas Y, Moilanen E, Salminen S. Probiotics in the management of atopic eczema. Clin Exp Allergy. 2000 Nov;30(11):1604-10. doi: 10.1046/j.1365-2222.2000.00943.x. PMID 11069570
- [Background] Kallio S, Kukkonen AK, Savilahti E, Kuitunen M. Perinatal probiotic intervention prevented allergic disease in a Caesarean-delivered subgroup at 13-year follow-up. Clin Exp Allergy. 2019 Apr;49(4):506-515. doi: 10.1111/cea.13321. Epub 2018 Dec 18. PMID 30472801
- [Background] Kalliomaki M, Salminen S, Arvilommi H, Kero P, Koskinen P, Isolauri E. Probiotics in primary prevention of atopic disease: a randomised placebo-controlled trial. Lancet. 2001 Apr 7;357(9262):1076-9. doi: 10.1016/S0140-6736(00)04259-8. PMID 11297958
- [Background] Kalliomaki M, Salminen S, Poussa T, Arvilommi H, Isolauri E. Probiotics and prevention of atopic disease: 4-year follow-up of a randomised placebo-controlled trial. Lancet. 2003 May 31;361(9372):1869-71. doi: 10.1016/S0140-6736(03)13490-3. PMID 12788576
- [Background] Karav S, Casaburi G, Frese SA. Reduced colonic mucin degradation in breastfed infants colonized by Bifidobacterium longum subsp. infantis EVC001. FEBS Open Bio. 2018 Sep 17;8(10):1649-1657. doi: 10.1002/2211-5463.12516. eCollection 2018 Oct. PMID 30338216
- [Background] Kela.fi: Maternity, Paternity and Parental Allowances [Internet]. Helsinki (Finland): Kansaneläkelaitos - The Social Insurance Institution of Finland; [updated 2020 Jan 16; cited 2020 Apr 27]. Available from: https://www.kela.fi/web/en/parental-allowances.
- [Background] Kim JY, Kwon JH, Ahn SH, Lee SI, Han YS, Choi YO, Lee SY, Ahn KM, Ji GE. Effect of probiotic mix (Bifidobacterium bifidum, Bifidobacterium lactis, Lactobacillus acidophilus) in the primary prevention of eczema: a double-blind, randomized, placebo-controlled trial. Pediatr Allergy Immunol. 2010 Mar;21(2 Pt 2):e386-93. doi: 10.1111/j.1399-3038.2009.00958.x. Epub 2009 Oct 14. PMID 19840300
- [Background] Kim CH, Park J, Kim M. Gut microbiota-derived short-chain Fatty acids, T cells, and inflammation. Immune Netw. 2014 Dec;14(6):277-88. doi: 10.4110/in.2014.14.6.277. Epub 2014 Dec 22. PMID 25550694
- [Background] Kukkonen K, Savilahti E, Haahtela T, Juntunen-Backman K, Korpela R, Poussa T, Tuure T, Kuitunen M. Probiotics and prebiotic galacto-oligosaccharides in the prevention of allergic diseases: a randomized, double-blind, placebo-controlled trial. J Allergy Clin Immunol. 2007 Jan;119(1):192-8. doi: 10.1016/j.jaci.2006.09.009. Epub 2006 Oct 23. PMID 17208601
- [Background] Lee MJ, Kang MJ, Lee SY, Lee E, Kim K, Won S, Suh DI, Kim KW, Sheen YH, Ahn K, Kim BS, Hong SJ. Perturbations of gut microbiome genes in infants with atopic dermatitis according to feeding type. J Allergy Clin Immunol. 2018 Apr;141(4):1310-1319. doi: 10.1016/j.jaci.2017.11.045. Epub 2018 Jan 12. PMID 29339259
- [Background] Lee SY, Lee E, Park YM, Hong SJ. Microbiome in the Gut-Skin Axis in Atopic Dermatitis. Allergy Asthma Immunol Res. 2018 Jul;10(4):354-362. doi: 10.4168/aair.2018.10.4.354. PMID 29949831
- [Background] Leung DYM, Calatroni A, Zaramela LS, LeBeau PK, Dyjack N, Brar K, David G, Johnson K, Leung S, Ramirez-Gama M, Liang B, Rios C, Montgomery MT, Richers BN, Hall CF, Norquest KA, Jung J, Bronova I, Kreimer S, Talbot CC Jr, Crumrine D, Cole RN, Elias P, Zengler K, Seibold MA, Berdyshev E, Goleva E. The nonlesional skin surface distinguishes atopic dermatitis with food allergy as a unique endotype. Sci Transl Med. 2019 Feb 20;11(480):eaav2685. doi: 10.1126/scitranslmed.aav2685. PMID 30787169
- [Background] Lewis ZT, Mills DA. Differential Establishment of Bifidobacteria in the Breastfed Infant Gut. Nestle Nutr Inst Workshop Ser. 2017;88:149-159. doi: 10.1159/000455399. Epub 2017 Mar 27. PMID 28346936
- [Background] Lowe AJ, Leung DYM, Tang MLK, Su JC, Allen KJ. The skin as a target for prevention of the atopic march. Ann Allergy Asthma Immunol. 2018 Feb;120(2):145-151. doi: 10.1016/j.anai.2017.11.023. PMID 29413338
- [Background] Netea MG, Joosten LA, Latz E, Mills KH, Natoli G, Stunnenberg HG, O'Neill LA, Xavier RJ. Trained immunity: A program of innate immune memory in health and disease. Science. 2016 Apr 22;352(6284):aaf1098. doi: 10.1126/science.aaf1098. Epub 2016 Apr 21. PMID 27102489
- [Background] Nocerino R, De Filippis F, Cecere G, Marino A, Micillo M, Di Scala C, de Caro C, Calignano A, Bruno C, Paparo L, Iannicelli AM, Cosenza L, Maddalena Y, Della Gatta G, Coppola S, Carucci L, Ercolini D, Berni Canani R. The therapeutic efficacy of Bifidobacterium animalis subsp. lactis BB-12(R) in infant colic: A randomised, double blind, placebo-controlled trial. Aliment Pharmacol Ther. 2020 Jan;51(1):110-120. doi: 10.1111/apt.15561. Epub 2019 Dec 3. PMID 31797399
- [Background] Penders J, Gerhold K, Stobberingh EE, Thijs C, Zimmermann K, Lau S, Hamelmann E. Establishment of the intestinal microbiota and its role for atopic dermatitis in early childhood. J Allergy Clin Immunol. 2013 Sep;132(3):601-607.e8. doi: 10.1016/j.jaci.2013.05.043. Epub 2013 Jul 27. PMID 23900058
- [Background] Rajka G, Langeland T. Grading of the severity of atopic dermatitis. Acta Derm Venereol Suppl (Stockh). 1989;144:13-4. doi: 10.2340/000155551441314. PMID 2800895
- [Background] Rautava S, Kalliomaki M, Isolauri E. Probiotics during pregnancy and breast-feeding might confer immunomodulatory protection against atopic disease in the infant. J Allergy Clin Immunol. 2002 Jan;109(1):119-21. doi: 10.1067/mai.2002.120273. PMID 11799376
- [Background] Rautava S, Kainonen E, Salminen S, Isolauri E. Maternal probiotic supplementation during pregnancy and breast-feeding reduces the risk of eczema in the infant. J Allergy Clin Immunol. 2012 Dec;130(6):1355-60. doi: 10.1016/j.jaci.2012.09.003. Epub 2012 Oct 16. PMID 23083673
- [Background] Ruohtula T, de Goffau MC, Nieminen JK, Honkanen J, Siljander H, Hamalainen AM, Peet A, Tillmann V, Ilonen J, Niemela O, Welling GW, Knip M, Harmsen HJ, Vaarala O. Maturation of Gut Microbiota and Circulating Regulatory T Cells and Development of IgE Sensitization in Early Life. Front Immunol. 2019 Oct 23;10:2494. doi: 10.3389/fimmu.2019.02494. eCollection 2019. PMID 31749800
- [Background] Schmidt RM, Pilmann Laursen R, Bruun S, Larnkjaer A, Molgaard C, Michaelsen KF, Host A. Probiotics in late infancy reduce the incidence of eczema: A randomized controlled trial. Pediatr Allergy Immunol. 2019 May;30(3):335-340. doi: 10.1111/pai.13018. Epub 2019 Feb 21. PMID 30790361
- [Background] Smilowitz JT, Moya J, Breck MA, Cook C, Fineberg A, Angkustsiri K, Underwood MA. Safety and tolerability of Bifidobacterium longum subspecies infantis EVC001 supplementation in healthy term breastfed infants: a phase I clinical trial. BMC Pediatr. 2017 May 30;17(1):133. doi: 10.1186/s12887-017-0886-9. PMID 28558732
- [Background] Sullivan M, Silverberg NB. Current and emerging concepts in atopic dermatitis pathogenesis. Clin Dermatol. 2017 Jul-Aug;35(4):349-353. doi: 10.1016/j.clindermatol.2017.03.006. Epub 2017 Mar 23. PMID 28709564
- [Background] Szajewska H, Horvath A. Lactobacillus rhamnosus GG in the Primary Prevention of Eczema in Children: A Systematic Review and Meta-Analysis. Nutrients. 2018 Sep 18;10(9):1319. doi: 10.3390/nu10091319. PMID 30231505
- [Background] Tannock GW, Lee PS, Wong KH, Lawley B. Why Don't All Infants Have Bifidobacteria in Their Stool? Front Microbiol. 2016 May 31;7:834. doi: 10.3389/fmicb.2016.00834. eCollection 2016. No abstract available. PMID 27303402
- [Background] Taylor AL, Dunstan JA, Prescott SL. Probiotic supplementation for the first 6 months of life fails to reduce the risk of atopic dermatitis and increases the risk of allergen sensitization in high-risk children: a randomized controlled trial. J Allergy Clin Immunol. 2007 Jan;119(1):184-91. doi: 10.1016/j.jaci.2006.08.036. Epub 2006 Oct 13. PMID 17208600
- [Background] Torow N, Hornef MW. The Neonatal Window of Opportunity: Setting the Stage for Life-Long Host-Microbial Interaction and Immune Homeostasis. J Immunol. 2017 Jan 15;198(2):557-563. doi: 10.4049/jimmunol.1601253. PMID 28069750
- [Background] Underwood MA, German JB, Lebrilla CB, Mills DA. Bifidobacterium longum subspecies infantis: champion colonizer of the infant gut. Pediatr Res. 2015 Jan;77(1-2):229-35. doi: 10.1038/pr.2014.156. Epub 2014 Oct 10. PMID 25303277
- [Background] van der Meulen TA, Harmsen H, Bootsma H, Spijkervet F, Kroese F, Vissink A. The microbiome-systemic diseases connection. Oral Dis. 2016 Nov;22(8):719-734. doi: 10.1111/odi.12472. Epub 2016 Apr 26. PMID 26953630
- [Background] Stm.fi: Maternity and Child Health Clinics [Internet]. Helsinki (Finland): Ministry of Social Affairs and Health; [cited 2020 Apr 27]. Available from: https://stm.fi/en/maternity-and-child-health-clinics.
- [Background] Vatanen T, Kostic AD, d'Hennezel E, Siljander H, Franzosa EA, Yassour M, Kolde R, Vlamakis H, Arthur TD, Hamalainen AM, Peet A, Tillmann V, Uibo R, Mokurov S, Dorshakova N, Ilonen J, Virtanen SM, Szabo SJ, Porter JA, Lahdesmaki H, Huttenhower C, Gevers D, Cullen TW, Knip M; DIABIMMUNE Study Group; Xavier RJ. Variation in Microbiome LPS Immunogenicity Contributes to Autoimmunity in Humans. Cell. 2016 May 5;165(4):842-53. doi: 10.1016/j.cell.2016.04.007. Epub 2016 Apr 28. PMID 27133167
- [Background] Wadonda-Kabondo N, Sterne JA, Golding J, Kennedy CT, Archer CB, Dunnill MG; ALSPAC Study Team. Association of parental eczema, hayfever, and asthma with atopic dermatitis in infancy: birth cohort study. Arch Dis Child. 2004 Oct;89(10):917-21. doi: 10.1136/adc.2003.034033. PMID 15383434
- [Background] Wang H, Li Y, Feng X, Li Y, Wang W, Qiu C, Xu J, Yang Z, Li Z, Zhou Q, Yao K, Wang H, Li Y, Li D, Dai W, Zheng Y. Dysfunctional gut microbiota and relative co-abundance network in infantile eczema. Gut Pathog. 2016 Jul 22;8:36. doi: 10.1186/s13099-016-0118-0. eCollection 2016. PMID 27453732
- [Background] Wassmann A, Werfel T. Atopic eczema and food allergy. Chem Immunol Allergy. 2015;101:181-90. doi: 10.1159/000371701. Epub 2015 May 21. PMID 26022878
- [Background] Weidinger S, Beck LA, Bieber T, Kabashima K, Irvine AD. Atopic dermatitis. Nat Rev Dis Primers. 2018 Jun 21;4(1):1. doi: 10.1038/s41572-018-0001-z. PMID 29930242
- [Background] Wickens K, Black PN, Stanley TV, Mitchell E, Fitzharris P, Tannock GW, Purdie G, Crane J; Probiotic Study Group. A differential effect of 2 probiotics in the prevention of eczema and atopy: a double-blind, randomized, placebo-controlled trial. J Allergy Clin Immunol. 2008 Oct;122(4):788-794. doi: 10.1016/j.jaci.2008.07.011. Epub 2008 Aug 31. PMID 18762327
- [Background] Zeevenhooven J, Koppen IJ, Benninga MA. The New Rome IV Criteria for Functional Gastrointestinal Disorders in Infants and Toddlers. Pediatr Gastroenterol Hepatol Nutr. 2017 Mar;20(1):1-13. doi: 10.5223/pghn.2017.20.1.1. Epub 2017 Mar 27. PMID 28401050
- [Background] Zheng H, Liang H, Wang Y, Miao M, Shi T, Yang F, Liu E, Yuan W, Ji ZS, Li DK. Altered Gut Microbiota Composition Associated with Eczema in Infants. PLoS One. 2016 Nov 3;11(11):e0166026. doi: 10.1371/journal.pone.0166026. eCollection 2016. PMID 27812181
- [Background] Zimmermann P, Messina N, Mohn WW, Finlay BB, Curtis N. Association between the intestinal microbiota and allergic sensitization, eczema, and asthma: A systematic review. J Allergy Clin Immunol. 2019 Feb;143(2):467-485. doi: 10.1016/j.jaci.2018.09.025. Epub 2018 Dec 29. PMID 30600099
- [Background] Zuccotti G, Meneghin F, Aceti A, Barone G, Callegari ML, Di Mauro A, Fantini MP, Gori D, Indrio F, Maggio L, Morelli L, Corvaglia L; Italian Society of Neonatology. Probiotics for prevention of atopic diseases in infants: systematic review and meta-analysis. Allergy. 2015 Nov;70(11):1356-71. doi: 10.1111/all.12700. Epub 2015 Aug 13. PMID 26198702